CLINICAL TRIAL: NCT05569213
Title: Combining Deep Brain Stimulation (DBS) and Motor Evoked Potentials (MEP) to Map Activation Loci in the Human Corticospinal Tract
Brief Title: Deep Brain Stimulation (DBS) and Motor Evoked Potentials (MEP)
Acronym: DBS MEP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: HS25589
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-08

CONDITIONS: MEP Onset Latency
MeSH Terms: interventions — Evoked Potentials, Motor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- DBS latency/MEP latency: Each patient will serve as control and test. Control will be latency of hand MEP generated by DBS stimulation of the corticospinal tract. The test condition will be the latency of hand MEP generated by conventional MEP acquisition.
  Interventions: Diagnostic Test: motor evoked potentials

INTERVENTIONS:
Diagnostic Test: motor evoked potentials — see previous descriptions

SUMMARY:
MEP onset latencies from the hand muscle using two different stimulus methods will be compared from each study participant. Conventional MEP data will be collected prior to skin incision. Following the DBS insertion hand muscle evoked responses will be generated via the DBS electrode. A hand held DBS programmer will be connected to the proximal end of the implanted DBS for delivery of electrical stimuli. Stimulus intensity will be adjusted until a hand muscle evoked potential is registered from the same recording electrodes used for the conventional MEP acquisition. A STN-implanted electrode can produce hand muscle responses due to it's close proximity to the motor fibres of the internal capsule. When the conventional and DBS-induced hand muscle responses have been acquired the study data objectives have been met. Data will be analyzed off-line.

DETAILED DESCRIPTION:
Purpose: Hand muscle MEP generated via the DBS electrode will provide an onset latency standard from which we can compare conventional MEP from the same hand muscles. It is critical for validation of conventional MEP to know where in the brain the motor pathway is being stimulated. This will avoid false negative MEP test results.

Objectives: We will measure the onset latencies from hand muscle MEP generated via the DBS electrode as well as using conventional MEP methods. The DBS onset latency data will provide a known anatomical standard to compare with conventional hand MEP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients scheduled for DBS surgery under general anesthesia; age 35-75 years; no history of stroke or peripheral nerve disease

Exclusion Criteria:

* peripheral nerve disease (e.g. type I diabetes); demyelinating disease (e.g. multiple sclerosis); previous stroke; allergy to propofol based anesthesia

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patient population will be those diagnosed with medically refractory Parkinson's Disease or Essential tremor and scheduled for DBS surgery.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Combining deep brain stimulation (DBS) and motor evoked potentials (MEP) to map activation loci in the human corticospinal tract | 12 months
  onset latency of motor evoked potentials

CONTACTS AND LOCATIONS:
Overall Officials: Marshall F Wilkinson, PhD, Principal Investigator — University of Manitoba

IPD SHARING:
Plan to Share IPD: Undecided
onset latencies derived from conventional and DBS-induced MEP will be available upon study completion